CLINICAL TRIAL: NCT06187675
Title: A Participant Choice Approach to Improve Adherence and Investigate Pregnancy Outcomes to Lifestyle Interventions
Brief Title: A Nutrition and Exercise Lifestyle Intervention Program Participant Choice Approach
Acronym: NELIP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Michelle Mottola, Principal Investigator, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 123317
Record Dates: First submitted 2023-11-30; First posted 2024-01-02 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Lifestyle, Healthy; Pregnancy Related; Adherence, Treatment; Nutrition, Healthy; Weight Gain, Maternal
Keywords: pregnancy; lifestyle; nutrition; exercise; adherence
MeSH Terms: conditions — Treatment Adherence and Compliance; Gestational Weight Gain; Motor Activity | interventions — Nutritional Status

STUDY DESIGN:
Intervention Model Description: pseudo randomized yoked design
Who Masked: Outcomes Assessor
Masking Description: data analysis will be analysed blinded to group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Choice (Active Comparator): Participants will be given a choice of 3 strategies; Group A - they receive both nutrition and exercise components simultaneously, Group B - they receive the nutrition component first followed by introduction of the exercise component sequentially, or Group C - they receive the exercise component first followed by introduction of the nutrition component sequentially.
  Interventions: Behavioral: Nutrition and Exercise Lifestyle Intervention Program
- No choice (Experimental): Participants will be yoked (matched) to a participant in the Choice group and they receive the same strategy as the person with a choice.
  Interventions: Behavioral: Nutrition and Exercise Lifestyle Intervention Program

INTERVENTIONS:
Behavioral: Nutrition and Exercise Lifestyle Intervention Program — Nutrition and Exercise components for pregnancy
  Other Names: NELIP

SUMMARY:
Interventions that target excessive gestational weight gain (EGWG) with nutrition and exercise behavior change struggle with low program adherence. The investigators recently examined adherence in a randomized controlled trial to a previously established lifestyle program called the Nutrition and Exercise Lifestyle Intervention Program (NELIP) and found that those individuals with high adherence to the program were more likely to prevent EGWG. Perhaps offering participants a choice to intervention strategies may improve adherence. The current research question is: What impact does participant choice have on adherence to the introduction of nutrition and exercise components during 3 intervention strategies offered to pregnant individuals compared to no choice and does choice maintain pregnancy health outcomes? The strategies are: Group A - introducing both the nutrition and exercise components simultaneous at baseline (12-18 weeks of pregnancy) that is followed to delivery (NELIP); Group B - introducing the nutrition component first and then at 25 weeks adding the exercise component; or Group C - starting with the exercise component first, followed with introducing the nutrition component at 25 weeks. Both Groups B and C follow the full NELIP from 25 weeks to delivery (final intervention measures will occur at 34-36 weeks gestation). Follow-up will occur at birth (6-18 hours), 2, 6 and 12 months post delivery.

DETAILED DESCRIPTION:
Investigators are using a pseudo randomized yoked design and will include two groups: choice of intervention strategy or no-choice. If the individual is randomized to no choice, then the next person would get a choice and the no choice person would be assigned to the group yoked (matched) to the person with a choice. Participants assigned to the choice group will choose one of three intervention strategies provided; either Group A (receiving both nutrition and exercise simultaneously), B (starting with nutrition and receiving exercise sequentially followed by nutrition starting at 25 weeks) or C (starting with nutrition first and then introducing exercise sequentially at 25 weeks). All groups will follow the full NELIP until delivery. Participants in the no-choice group will be yoked (matched) to a participant in the choice group and receive the strategy that their yoked counterparts chose.

Nutrition component of NELIP: This component is a modified gestational diabetic meal plan that has four general goals tailored to the participant: (1) to achieve approximately 2000 kcal of energy per day. The determination of the amount of kcal consumed per day will consider the participant's intake from the dietary assessment. There also must not be a restriction of calories that exceeds 30% of their total energy intake; (2) participants will consume approximately 200-250g/day of carbohydrates, accounting for approximately 40-55% of total energy intake. Carbohydrate intake will be distributed throughout three meals and four snacks daily. The nutritionist will educate participants about the importance of complex and low-glycemic index carbohydrates through the one-on-one session; (3) fat and protein intake will be approximately 30% and 20-30% of total energy intake, respectively; (4) achieve appropriate micronutrient and fluid intake for pregnancy. This will be monitored by a weekly 24 hour food intake record.

Exercise component of NELIP: This is a walking program that comprises of 1 weekly supervised session on a treadmill or outside and participants will be recommended to walk 2 to 3 additional times per week. The walking program will start at 25 minutes per session, 3 to 4 times weekly, and increase by 2 minutes per week until 40 minutes and then maintained until delivery. This will be monitored by a wrist monitoring device. The primary outcome is adherence measured weekly using a published adherence protocol using a point system. Secondary outcomes are participant satisfaction to the program and health outcomes: weekly weight gain, calculated EGWG, and pregnancy outcomes (birth weight length, infant anthropometrics, APGAR scores and delivery complications). At 2, 6 and 12 months of age the maternal-infant dyad will return to the lab and infant morphometric measurements recorded from birth will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* between 12 to 18 weeks of pregnancy
* a singleton fetus
* medically screened with the Get Active Questionnaire for Pregnancy to determine eligibility for participation in the exercise component

Exclusion Criteria:

* inability to walk
* serious medical problems
* high blood pressure
* uncontrolled chest pain
* uncontrolled symptomatic lung disease
* diabetes before pregnancy
* a history of recreational substance use disorder
* any contraindication to exercise
* enrolled in another clinical trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — All gender identities will be accepted as these individuals must be pregnant.
Enrollment: 120 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Adherence to the intervention strategy | Measured once per week from baseline (12-18 weeks gestation) to end of the intervention (34-36 weeks gestation)
  Percent of participants adherent to the strategies measured by a published Adherence Scale giving a score out of 3 for each component (nutrition and exercise).

SECONDARY OUTCOMES:
Participant satisfaction | Measured at 34-36 weeks of pregnancy at the end of the intervention
  Satisfaction Survey assessed on a 5-point Likert scale; ranging from 1 for very unsatisfied to 5 for very satisfied.
Gestational weight gain | Measured weekly from 12-18 weeks of pregnancy to 34-36 weeks of pregnancy
  Weight gained measured in kg and compared to the Institute of Medicine 2009 weight gain guidelines
Birth weight | Measured within 6 to 18 hours after delivery
  Birth weight (measured in kg)
Birth length | Measured within 6 to 18 hours after delivery
  Birth Length (measured in cms)
Birth circumferences | Measured within 6 to 18 hours after delivery
  Newborn circumferences (arm, forearm, thigh, leg, abdomen, chest, and head - measured in cm)
Birth skinfolds | Measured within 6 to 18 hours after delivery
  Newborn skinfolds (biceps, triceps, subscapular, suprailiac, anterior thigh - measured in mm)
Pregnancy outcome | Measured within 6 to 18 hours after delivery
  APGAR scores (measured out of 10 at 1 minutes and 5 minutes after birth)
Pregnancy complications | Measured within 6 to 18 hours after delivery
  Pregnancy complications (recorded)
Postpartum body weight | 2, 6 and 12 months after birth
  Participant body weight (measured in kg)
Follow-up Infant weight | 2, 6 and 12 months after birth
  Infant weight (measured in kg)
Follow-up Infant length | 2, 6 and 12 months after birth
  Infant length (measured in cm)
Follow-up Infant Girths | 2, 6 and 12 months after birth
  Infant circumferences (arm, forearm, thigh, leg, abdomen, chest, head - measured in cm)
Follow-up Infant adiposity | 2, 6 and 12 months after birth
  Infant skinfold measurements (biceps, triceps, subscapular, suprailiac, anterior thigh - measured in mm)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle F Mottola, PhD, Principal Investigator — Western University
Locations (1):
- Exercise and Pregnancy Lab, 2245, 3-M Centre - University of Western Ontario, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
deidentified data may be shared after publication
Supporting Information: Study Protocol
Time Frame: After completion of the study and after publication
Access Criteria: Access with be determined by the principal investigator once the reasons for data acquisition are given

REFERENCES:
- [Background] Nagpal TS, Prapavessis H, Campbell CG, de Vrijer B, Bgeginski R, Hosein K, Paplinskie S, Manley M, Mottola MF. Sequential Introduction of Exercise First Followed by Nutrition Improves Program Adherence During Pregnancy: a Randomized Controlled Trial. Int J Behav Med. 2020 Feb;27(1):108-118. doi: 10.1007/s12529-019-09840-0. PMID 31872340
- [Background] Nagpal TS, Prapavessis H, Campbell C, Mottola MF. Measuring Adherence to a Nutrition and Exercise Lifestyle Intervention: Is Program Adherence Related to Excessive Gestational Weight Gain? Behav Anal Pract. 2017 May 17;10(4):347-354. doi: 10.1007/s40617-017-0189-5. eCollection 2017 Dec. PMID 29214130
- [Background] Mottola MF, Giroux I, Gratton R, Hammond JA, Hanley A, Harris S, McManus R, Davenport MH, Sopper MM. Nutrition and exercise prevent excess weight gain in overweight pregnant women. Med Sci Sports Exerc. 2010 Feb;42(2):265-72. doi: 10.1249/MSS.0b013e3181b5419a. PMID 20083959
- See also: Exercise and Pregnancy Laboratory Website — http://www.uwo.ca/fhs/EPL